CLINICAL TRIAL: NCT06420310
Title: Prevalence of Preclinical and Prodromal Parkinson´s Disease in Subjects Exposed to Pesticides
Brief Title: Pesticides and Parkinson´s Disease
Acronym: Pest-PD
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario de Burgos (Other)
Responsible Party: Principal Investigator, Esther Cubo, MD, PhD, Hospital Universitario de Burgos
Other Study IDs: GRS 2682/A1/2023
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Pesticide-Induced Parkinsonism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood samples from cases and controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Subjects exposed to pesticides
  Interventions: Other: exposure to pesticides
- Controls: Subjects without any exposure to pesticides
  Interventions: Other: exposure to pesticides

INTERVENTIONS:
Other: exposure to pesticides — based on work exposures to pesticides

SUMMARY:
The aim of this project is to study whether people exposed to pesticides have a higher risk of developing PD. We will perform an epidemiological study determining the presence of pesticides in urine and comparing signs traditionally associated with PD in early forms.

DETAILED DESCRIPTION:
Within different risk factors, pesticide exposure increases the risk of developing Parkinson's disease (PD) through epigenetic mechanisms by modifying the expression of genes related to PD and secondary mitochondrial dysfunction.We will conduct a cross-sectional prevalence study with cases (exposed to pesticides) and controls (not exposed to pesticides), randomly selecting 130 individuals in each group. Pesticide exposure will be determined through questionnaires.We will study the prevalence of preclinical and prodromal PD based on pesticide exposure, stratified by age and gender in the exposed, and non-exposed groups. Preclinical and prodromal PD will be assessed using: biological biomarkers and prodromal PD signs. Multivariate analyses will be employed to determine the risk of presenting early PD, adjusting for different clinical covariates. The results of this study will allow us to understand the early mechanisms associated with neurodegeneration and pesticides exposure.

ELIGIBILITY:
Inclusion Criteria:

* Farmers exposed to pesticides for cases
* No work exposure to pesticides for controls

Exclusion Criteria:

* Subjects without signed consent form
* Neurological significant conditions

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects not diagnosed with PD living in Burgos region
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Prodromal PD | over the last year
  Early non motor symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No